CLINICAL TRIAL: NCT05622162
Title: Phase III Multicentre Prospective Comparative Study of Detection Rate of 18F-JK-PSMA-7 and of 18F-fluorocholine in Patients With Biochemical Recurrence of Prostate Cancer After Previous Treatment With Curative Intent
Brief Title: Prospective Comparative Study for Patients With Biochemical Recurrence Prostate Cancer Detecting by 18F-JK-PSMA-7
Acronym: MIP7
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ITEL Telecomunicazioni Srl (Industry)
Collaborators: Advice Pharma Group srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2021-005993-24
Record Dates: First submitted 2022-11-09; First posted 2022-11-18 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer; 18F- Fluorocholine; PSMA PET; Radiotherapy; Prostatectomy; Tumor of Prostate
Keywords: Prostate Cancer; Prostatectomy; diagnostic radiopharmaceutical; PET; CT; PSA; Biochemical Recurrence; 18F- Fluorocholine; 18F-JK-PSMA-7; PSMA; Standard of truth
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 18F-JK-PSMA-7; fluorocholine

STUDY DESIGN:
Intervention Model Description: Prospective, multicentric, comparative (controlled), phase III study of diagnostic performance with blind reading and standard of truth.
Masking Description: The blind readers of PET/CT examinations with Investigational product (18F-JK-PSMA-7) and with Comparator (18F-fluorocholine) will be blinded to any clinical data of patient.
  The analysis of images obtained with IMP (18F-JK-PSMA-7) and with Comparator (18F-fluorocholine) will be performed by two independent off-site experts blinded to any patient´s clinical data, using the defined grid (Appendix I). Discrepancies between results of the two observers will be recorded by the clinical manager and a consensus reading with third expert will be organized. This reading will be used for determination of imaging performances.
  Wash-out period of at least one month is ensured between reading of examinations with Investigational product (18F-JK-PSMA-7) and with Comparator (18F-Fluorocholine) for each blind reader.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional and Comparator (Experimental): The subject participation in the study consists from performing of one non-contrast enhanced PET/CT with Investigational Product (18F-JK-PSMA-7) and of one PET/CT with Comparator (18F-Fluorocholine) This sequence of administration is established in advance as the organizational model, linked to the availability and management of the radiopharmaceutical, not allow to perform a randomization.
  Interventions: Drug: Radiopharmaceutical 18F-JK-PSMA-7; Drug: Radiopharmaceutical 18F-Fluorocholine

INTERVENTIONS:
Drug: Radiopharmaceutical 18F-JK-PSMA-7 — The Investigational product 18F-JK-PSMA-7 is a diagnostic radiopharmaceutical for use with positron emission tomography.
  18F-JK-PSMA-7 is administered as direct intravenous injection. One single administration of 2-4 MBq/kg of 18F-JK-PSMA-7 is scheduled in each patient included in this study.
  Other Names: 18F-JK-PSMA-7
Drug: Radiopharmaceutical 18F-Fluorocholine — The active substance of Comparator is 18F-Fluorocholine. The Comparator will be a 18F-Fluorocholine with a Marketing Authorisation in Italy that will be used in compliance with its Summary of Product Characteristics (SmPC).
  18F-Fluorocholine is administrated as direct intravenous injection. One single administration of 18F-Fluorocholine is scheduled in each patient included in this study.
  Other Names: 18F-Fluorocholine

SUMMARY:
The present study in patients with Prostate cancer and biochemical failure after surgery and/or radical-postoperative Radio Therapy (RT) will evaluate if PET/CT with 18F-JK-PSMA-7 compared to PET-CT 18F-Choline is able to identify the early pattern of biochemical recurrence and/or metastatic sites, so that the patient could be better managed, with a benefit in survival.

DETAILED DESCRIPTION:
Investigational Product:

The investigational product in this study is 18F-JK-PSMA-7, a fluorine-18 labelled ligand binding specifically to prostate specific membrane antigen (PSMA).

The investigational product 18F-JK-PSMA-7 is a diagnostic radiopharmaceutical for use with positron emission tomography (PET).

The active substance of the diagnostic radiopharmaceutical product is 18F-JK-PSMA-7.

Fluorine (F) decays to stable oxygen (O) with a half-life of 110 minutes by emitting a positronic radiation of maximum energy of 634 keV, followed by photonic annihilation radiations of 511 keV.

The investigational product 18F-JK-PSMA-7 is a newly developed F-labelled PET tracer for functional imaging of PSMA expression.

PSMA is a transmembrane glycoprotein that is expressed in a variety of cells and is characterized by its overexpression in Prostate Cancer. The overexpression of PSMA has been observed both in primary Prostate Cancer as well as in metastatic lesions.

The active substance of Comparator is 18F-Fluorocholine. The Comparator will be a 18F-Fluorocholine with a Marketing Authorization in Italy that will be used in compliance with its Summary of Product Characteristics (SmPC).

18F-Fluorocholine is administrated as direct intravenous injection. One single administration of 18F-Fluorocholine is scheduled in each patient included in this study.

The analysis of images obtained with IMP (18F-JK-PSMA-7) and with Comparator (18F-fluorocholine) will be performed by two independent off site experts blinded to any patient´s clinical data, using the defined grid. Discrepancies between results of the two observers will be recorded by the clinical manager and a consensus reading with third expert will be organized. This reading will be used for determination of imaging performances.

Study duration.

* The study starts with a screening visit (-1), in which the medical history is collected, then a PET/TC examination (T0) is performed. The first examination will be performed with IMP.
* Whitin one month, a second PET-TC is performed using the Comparator, the other radiotracer (T1). Only for IMP are requested additional test of the tolerability (blood pressure, heart rate and inspection of injection site). The result of PET is analyzed by onsite reader, then by two blind out-site readers (blind to any clinical patient's data). A maximum wash-out period of 1 month is requested between the first and second reading performed by blind readers, in order to avoid that the reading can be affected by the knowledge of the first PET/TC examination.
* After 3 (T2) and 6 (T3) months from the last PET/TC examination (T1) a follow up visit will be performed in order to collect all the information related to procedures (treatments and/or examinations) performed by the patient according to clinical practices.
* After last visit and last patient (LVLP) of each site, the Assessment of Standard of Truth (SOT is established by a panel of expert blinded to result of PET/CT examination on the base of clinical data available in eCRF) and Performance evaluation will be performed (the Performance evaluation is an automatic determination); the estimated time for these activities is 6 months.
* In conclusion, each patient will be involved in the study about 7 months.

Two PET-TC will perform within one month of distance according to the following order: first the IMP than the Comparator.

This sequence of administration is established in advance as the organizational model, linked to the availability and management of the radiopharmaceutical, not allow to perform a randomization.

Risk and Benefits. The potential benefit from performing 18F-JK-PSMA-7 PET/CT in addition to PET/CT with Comparator in patients with biochemical recurrence of Prostate Cancer after primary treatment with curative intent consists from expected earlier and more sensitive localization of sites of recurrent disease than with 18F-Fluorocholine PET/CT which is currently the only one diagnostic radiopharmaceutical for use with PET approved for localization of lesions of recurrent Prostate Cancer. The early recognition of the disease resumption can allow the use of targeted treatments that can postpone the use of hormone therapy or, in case of metastatic disease, the use of systemic treatment.

In conclusion, the benefit / risk ratio for the patients involved is widely considered positive.

Primary objective. To show in an independent assessment by two readers blinded to clinical data the superiority of 18F-JK-PSMA-7 over 18F-Fluorocholine in patient-based detection rate of recurrent Prostate Cancer in patients with confirmed biochemical recurrence after treatment with curative intention.

Based on available bibliographic data we hypothesize that the detection rate of 18F-JKPSMA-7 is at least 20% higher than that of 18F-Fluorocholine.

Secondary objective.

* To evaluate the site-based sensitivity and specificity of 18F-JK-PSMA-7 and of 18F-Fluorocholine PET/CT for recurrent Prostate Cancer;
* To evaluate the frequency of change of actual therapeutic management motivated by result of 18F-JK-PSMA-7 and by 18F-Fluorocholine PET/CT in comparison with initially scheduled therapeutic management;
* To evaluate the discordance rate in 18F-JK-PSMA-7 and in 18F-Fluorocholine PET/CT reading among two blinded readers;
* To evaluate the safety profile of 18F-JK-PSMA-7 and of 18F-Fluorocholine.

Primary endpoints

• The patient-based detection rate of 18F-JK-PSMA-7 and of 18F-Fluorocholine PET/CT as a result of consensus of blind reading using an expert panel as a SOT. The eventual major discordance of results of blind readings will be solved by third reader blinded to results of previous blind readings. In particular, the study hypohesizes a 20% diagnostic superiority of 18F-JK-PSMA-7 versus 18F- Fluorocholine. The primary objective of the study is the identification of the possible best diagnostic rate of 18F-JK-PSMA-7 versus 18F- Fluorocholine in identiofying the reccurance of prostatic disesase in patients previusly subjected to prostectomy. Furthemore, the aim of the study is to evaluate the diagnostic accuracy of 18F-JK-PSMA-7 versus 18F- Fluorocholine even for low PSA levels, where the 18F- Fluorocholine is considered to be insensitive in these conditions..

Secondary endpoints

* The site-based sensitivity and specificity of 18F-JK-PSMA-7 and of 18F-Fluorocholine PET/CT of foci of recurrent Prostate Cancer;
* The change of actual therapeutic management motivated by result of 18F-JK-PSMA-7 and of 18F-Fluorocholine PET/CT in comparison with initially scheduled therapeutic management;
* The discordance rate in 18F-JK-PSMA-7 and in 18F-Fluorocholine PET/CT reading among two blinded readers;
* The adverse events or reactions related with use of 18F-JK-PSMA-7 and with use of 18F-fluorocholine

Statistical analysis The usual descriptive statistics, sample size (n), mean, standard deviation, median and range will be provided for the quantitative variables as well as the actual and percentage for each category of the qualitative variables.

Proportions comparisons: Chi-square test (X2), or Fisher test (F) when appropriated, are the tests of choice. If tests corrections are performed, estimations for both the corrected and the non-corrected tests will be provided.

To evaluate the study hypothesis, the 95% confidence interval (CI) of the difference between the 18F-JK-PSMA-7 and 18F-Fluorocholine positive results will be evaluated as follows:

1. the proportion of positives of the two tests will be said to be different if the CI of the difference does not include the number zero and consequently considered different at 5% statistical significance level;
2. the extent in which the two tests differ will be reported using the width of the CI;
3. the difference will be said to be clinically significant if the lower bound of the CI does not include the value 20% (the superiority hypothesis).

Sample Size The sample size was calculated on the basis of the diagnostic performances of the 18F-Fluorocholine PET/CT present in the literature. Three subgroups were identified.

Groups are identified by PSA ng/mL level. A sample size calculation was performed for each subgroup, considering the performance of the PET-18F-Fluorocholine and of the PET-18F-JK-PSMA-7 in that subgroup and computing the sample size adequate for testing the one-side hypothesis H0: pPSMA = pPSMA - superiority margin versus H1: pPSMA > pPSMA - superiority margin where: pPSMA is supposed to be 0.8 in the first subgroup of PSA, 0.95 in the second subgroup and 0.98 in the third one; the superiority margin is equal to 0.2 in the first two subgroup of PSA and 0.15 in the third one.

So, with an α=0.05 and a power (1-β) = 0.80:

* in the subgroup A, 33 patients are needed in order to test H0: pPSMA=0.6 (0.8-0.2) vs H1: pPSMA>0.6;
* in the subgroup B, 21 patients are needed in order to test H0: pPSMA=0.75 (0.95-0.2) vs H1: pPSMA>0.75;
* in the subgroup C, 25 patients are needed in order to test H0: pPSMA=0.83 (0.98-0.15) vs H1: pPSMA>0.83.

The resulting sample size is 79 patients. These resulting was incremented considering a dropout rate of 25%, obtaining 79/0.75 = 106 patients to be enrolled.

The sponsor is responsible for implementing and maintaining quality assurance and quality control systems to ensure that trials are conducted, and data are generated, documented (recorded), and reported in compliance with the protocol, GCP, and the applicable regulatory requirements.

The Sponsor is responsible for securing agreement from all involved parties to ensure direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the Sponsor, and inspection by domestic and foreign regulatory authorities.

Quality control should be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly.

Agreements, made by the Sponsor with the investigator/institution and any other parties involved with the clinical trial, should be in writing, in protocol or in a separate agreement.

This study will be performed in accordance with the principles stated in the Declaration of Helsinki and subsequent amendments and in accordance with the Good Clinical Practice Guideline (CPMP/ICH/135/95).

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of prostate malignancy
2. Patient must have had their primary PCa treated with surgery and/or radiation therapy; salvage radiation to the prostate bed or pelvis is allowed
3. Patient must be ≥ 18 years of age
4. Patient must have an Eastern Cooperative Oncology Group performance status ≤ 2
5. For patients treated with radical prostatectomy: arise of PSA ≥ 0.2 ng/mL (performed in the last month) or a rise of 2 ng/mL or more above the nadir PSA after definitive radiation therapy defined by two subsequent PSA assessments performed over a 3-month period in the same laboratory
6. Absence of any of the exclusion criteria
7. Signed informed consent

Exclusion Criteria:

1. Absence of any of the inclusion criteria;
2. More than 3 years of androgen deprivation therapy (ADT), with less than 3 months from the last treatment
3. Spinal cord compression or impending spinal cord compression
4. Receipt of any other investigational agents in the previous 3 months
5. Inability to lie flat during or tolerate PET/CT
6. Hypersensitivity to active substance or any of excipients of Investigational Medicinal Product or Comparator
7. Life expectancy <6 months
8. ECOG performance status >2
9. Refusal to sign informed consent
10. Participation in a concurrent clinical trial
11. Concomitant active malignancy
12. Subject deprived of its freedom by administrative or legal decision or who is under guardianship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Detection rate of 18F-JK-PSMA-7 PET/CT | 1 Months
  To evaluate the diagnostic accuracy of 18F-JK-PSMA-7 versus 18F- Fluorocholine even for low PSA levels, where the 18F- Fluorocholine is considered to be insensitive in these conditions.
  Hypothesis: a 20% diagnostic superiority of 18F-JK-PSMA-7 versus 18F- Fluorocholine.

SECONDARY OUTCOMES:
Evaluation of the safety profile of 18F-JK-PSMA-7 | 6 months
  This outcome will be evaluated by the adverse events or reactions related with use of 18F-JK-PSMA-7 and with use of 18F-fluorocholine.
  Detected by the clinicians during the clinical study.
Evaluation of the discordance rate between IMP and Comparator | 1 month
  The discordance rate in 18F-JK-PSMA-7 and 18F-Fluorocholine PET/CT reading among two blinded operators will be calculated as a proportion of site-based and patient-based discordant findings out of all site-based and patient-based findings. Only the frequency of major discordances will be assessed (i.e. discordance in terms of malignant and benign character of lesions/sites or discordance in terms of patient-based positivity or negativity for recurrent PCa).
Influence of 18F-JK-PSMA-7 in the therapeutic management decision | 6 months
  The frequency of change of actual therapeutic management motivated by result of 18F-JK-PSMA-7 PET/CT in comparison with initially scheduled therapeutic management will be calculated by comparing initially scheduled therapeutic management and actual therapeutic management decided after 18F-JK-PSMA-7 and of 18F-Fluorocholine PET/CT.
Evaluation of sensitivity of 18F-JK-PSMA-7 | 6 months
  The site-based sensitivity of 18F-JK-PSMA-7 and of 18F-Fluorocholine PET/CT for localisation of foci of recurrent PCa will be calculated by comparison of results of blind reading with SOT.
Evaluation of specificity of 18F-JK-PSMA-7 | 6 months
  The site-based sensitivity and specificity of 18F-JK-PSMA-7 and of 18F-Fluorocholine PET/CT for localisation of foci of recurrent PCa will be calculated by comparison of results of blind reading with SOT.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - I.R.S.T. Srl Irccs, Meldola, Forlì-Cesena
  - Ospedale Classificato Sacro Cuore - Don Calabria, Negrar, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galgano SJ, Valentin R, McConathy J. Role of PET imaging for biochemical recurrence following primary treatment for prostate cancer. Transl Androl Urol. 2018 Sep;7(Suppl 4):S462-S476. doi: 10.21037/tau.2018.06.09. PMID 30363475
- [Result] Afshar-Oromieh A, Avtzi E, Giesel FL, Holland-Letz T, Linhart HG, Eder M, Eisenhut M, Boxler S, Hadaschik BA, Kratochwil C, Weichert W, Kopka K, Debus J, Haberkorn U. The diagnostic value of PET/CT imaging with the (68)Ga-labelled PSMA ligand HBED-CC in the diagnosis of recurrent prostate cancer. Eur J Nucl Med Mol Imaging. 2015 Feb;42(2):197-209. doi: 10.1007/s00259-014-2949-6. Epub 2014 Nov 20. PMID 25411132
- [Result] Afshar-Oromieh A, Zechmann CM, Malcher A, Eder M, Eisenhut M, Linhart HG, Holland-Letz T, Hadaschik BA, Giesel FL, Debus J, Haberkorn U. Comparison of PET imaging with a (68)Ga-labelled PSMA ligand and (18)F-choline-based PET/CT for the diagnosis of recurrent prostate cancer. Eur J Nucl Med Mol Imaging. 2014 Jan;41(1):11-20. doi: 10.1007/s00259-013-2525-5. Epub 2013 Sep 27. PMID 24072344
- [Result] Bauman G, Belhocine T, Kovacs M, Ward A, Beheshti M, Rachinsky I. 18F-fluorocholine for prostate cancer imaging: a systematic review of the literature. Prostate Cancer Prostatic Dis. 2012 Mar;15(1):45-55. doi: 10.1038/pcan.2011.35. Epub 2011 Aug 16. PMID 21844889
- [Result] Beheshti M, Haim S, Zakavi R, Steinmair M, Waldenberger P, Kunit T, Nader M, Langsteger W, Loidl W. Impact of 18F-choline PET/CT in prostate cancer patients with biochemical recurrence: influence of androgen deprivation therapy and correlation with PSA kinetics. J Nucl Med. 2013 Jun;54(6):833-40. doi: 10.2967/jnumed.112.110148. Epub 2013 Apr 4. PMID 23559588
- [Result] Castellucci P, Fanti S. Prostate cancer: Identifying sites of recurrence with choline-PET-CT imaging. Nat Rev Urol. 2015 Mar;12(3):134-5. doi: 10.1038/nrurol.2014.321. Epub 2014 Dec 2. No abstract available. PMID 25447835
- [Result] Decaestecker K, De Meerleer G, Lambert B, Delrue L, Fonteyne V, Claeys T, De Vos F, Huysse W, Hautekiet A, Maes G, Ost P. Repeated stereotactic body radiotherapy for oligometastatic prostate cancer recurrence. Radiat Oncol. 2014 Jun 12;9:135. doi: 10.1186/1748-717X-9-135. PMID 24920079
- [Result] Dietlein F, Hohberg M, Kobe C, Zlatopolskiy BD, Krapf P, Endepols H, Tager P, Hammes J, Heidenreich A, Neumaier B, Drzezga A, Dietlein M. An 18F-Labeled PSMA Ligand for PET/CT of Prostate Cancer: First-in-Humans Observational Study and Clinical Experience with 18F-JK-PSMA-7 During the First Year of Application. J Nucl Med. 2020 Feb;61(2):202-209. doi: 10.2967/jnumed.119.229542. Epub 2019 Jul 19. PMID 31324713
- [Result] Eiber M, Kroenke M, Wurzer A, Ulbrich L, Jooss L, Maurer T, Horn T, Schiller K, Langbein T, Buschner G, Wester HJ, Weber W. 18F-rhPSMA-7 PET for the Detection of Biochemical Recurrence of Prostate Cancer After Radical Prostatectomy. J Nucl Med. 2020 May;61(5):696-701. doi: 10.2967/jnumed.119.234914. Epub 2019 Dec 13. PMID 31836682
- [Result] Fuccio C, Rubello D, Castellucci P, Marzola MC, Fanti S. Choline PET/CT for prostate cancer: main clinical applications. Eur J Radiol. 2011 Nov;80(2):e50-6. doi: 10.1016/j.ejrad.2010.07.023. Epub 2010 Aug 25. PMID 20800404
- [Result] Giovacchini G, Giovannini E, Borso E, Lazzeri P, Riondato M, Leoncini R, Duce V, Conti E, Picchio M, Ciarmiello A. Sensitivity of fluorine-18-fluoromethylcholine PET/CT to prostate-specific antigen over different plasma levels: a retrospective study in a cohort of 192 patients with prostate cancer. Nucl Med Commun. 2019 Mar;40(3):258-263. doi: 10.1097/MNM.0000000000000959. PMID 30507748
- [Result] Heidenreich A, Bastian PJ, Bellmunt J, Bolla M, Joniau S, van der Kwast T, Mason M, Matveev V, Wiegel T, Zattoni F, Mottet N; European Association of Urology. EAU guidelines on prostate cancer. part 1: screening, diagnosis, and local treatment with curative intent-update 2013. Eur Urol. 2014 Jan;65(1):124-37. doi: 10.1016/j.eururo.2013.09.046. Epub 2013 Oct 6. PMID 24207135
- [Result] Kroenke M, Wurzer A, Schwamborn K, Ulbrich L, Jooss L, Maurer T, Horn T, Rauscher I, Haller B, Herz M, Wester HJ, Weber WA, Eiber M. Histologically Confirmed Diagnostic Efficacy of 18F-rhPSMA-7 PET for N-Staging of Patients with Primary High-Risk Prostate Cancer. J Nucl Med. 2020 May;61(5):710-715. doi: 10.2967/jnumed.119.234906. Epub 2019 Dec 13. PMID 31836681
- [Result] Mamede M, Ceci F, Castellucci P, Schiavina R, Fuccio C, Nanni C, Brunocilla E, Fantini L, Costa S, Ferretti A, Colletti PM, Rubello D, Fanti S. The role of 11C-choline PET imaging in the early detection of recurrence in surgically treated prostate cancer patients with very low PSA level <0.5 ng/mL. Clin Nucl Med. 2013 Sep;38(9):e342-5. doi: 10.1097/RLU.0b013e31829af913. PMID 23797218
- [Result] Menard C, Iupati D, Publicover J, Lee J, Abed J, O'Leary G, Simeonov A, Foltz WD, Milosevic M, Catton C, Morton G, Bristow R, Bayley A, Atenafu EG, Evans AJ, Jaffray DA, Chung P, Brock KK, Haider MA. MR-guided prostate biopsy for planning of focal salvage after radiation therapy. Radiology. 2015 Jan;274(1):181-91. doi: 10.1148/radiol.14122681. Epub 2014 Sep 8. PMID 25203127
- [Result] Natarajan A, Agrawal A, Murthy V, Bakshi G, Joshi A, Purandare N, Shah S, Puranik A, Rangarajan V. Initial experience of Ga-68 prostate-specific membrane antigen positron emission tomography/computed tomography imaging in evaluation of biochemical recurrence in prostate cancer patients. World J Nucl Med. 2019 Jul-Sep;18(3):244-250. doi: 10.4103/wjnm.WJNM_47_18. PMID 31516367
- [Result] Grummet J, Eggener S. Re: NCCN Prostate Cancer Guidelines Version 1.2022 - September 10, 2021. Eur Urol. 2022 Feb;81(2):218. doi: 10.1016/j.eururo.2021.11.025. Epub 2021 Dec 9. No abstract available. PMID 34895925
- [Result] Oh SW, Cheon GJ. Prostate-Specific Membrane Antigen PET Imaging in Prostate Cancer: Opportunities and Challenges. Korean J Radiol. 2018 Sep-Oct;19(5):819-831. doi: 10.3348/kjr.2018.19.5.819. Epub 2018 Aug 6. PMID 30174470
- [Result] Perera M, Papa N, Christidis D, Wetherell D, Hofman MS, Murphy DG, Bolton D, Lawrentschuk N. Sensitivity, Specificity, and Predictors of Positive 68Ga-Prostate-specific Membrane Antigen Positron Emission Tomography in Advanced Prostate Cancer: A Systematic Review and Meta-analysis. Eur Urol. 2016 Dec;70(6):926-937. doi: 10.1016/j.eururo.2016.06.021. Epub 2016 Jun 28. PMID 27363387
- [Result] Perks J, Benedict S. MO-F-BRCD-02: SBRT (Part 2): Physics and Quality Assurance Updates. Med Phys. 2012 Jun;39(6Part21):3873. doi: 10.1118/1.4735813. PMID 28518227
- [Result] Rahbar K, Afshar-Oromieh A, Seifert R, Wagner S, Schafers M, Bogemann M, Weckesser M. Diagnostic performance of 18F-PSMA-1007 PET/CT in patients with biochemical recurrent prostate cancer. Eur J Nucl Med Mol Imaging. 2018 Nov;45(12):2055-2061. doi: 10.1007/s00259-018-4089-x. Epub 2018 Jul 20. PMID 30027419
- [Result] Rajasekaran AK, Anilkumar G, Christiansen JJ. Is prostate-specific membrane antigen a multifunctional protein? Am J Physiol Cell Physiol. 2005 May;288(5):C975-81. doi: 10.1152/ajpcell.00506.2004. PMID 15840561
- [Result] Samper Ots P, Luis Cardo A, Vallejo Ocana C, Cabeza Rodriguez MA, Glaria Enriquez LA, Couselo Paniagua ML, Olivera Vegas J. Diagnostic performance of 18F-choline PET-CT in prostate cancer. Clin Transl Oncol. 2019 Jun;21(6):766-773. doi: 10.1007/s12094-018-1985-2. Epub 2018 Nov 17. PMID 30448957
- [Result] Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: Updated guidelines for reporting parallel group randomised trials. J Pharmacol Pharmacother. 2010 Jul;1(2):100-7. doi: 10.4103/0976-500X.72352. No abstract available. PMID 21350618
- [Result] Zlatopolskiy BD, Endepols H, Krapf P, Guliyev M, Urusova EA, Richarz R, Hohberg M, Dietlein M, Drzezga A, Neumaier B. Discovery of 18F-JK-PSMA-7, a PET Probe for the Detection of Small PSMA-Positive Lesions. J Nucl Med. 2019 Jun;60(6):817-823. doi: 10.2967/jnumed.118.218495. Epub 2018 Nov 2. PMID 30389823
- See also: Farmacopea Europea X edizione — https://www.certifico.com/chemicals/legislazione-chemicals/10448-decreto-9-febbraio-2020-10-edizione-della-farmacopea-europea